CLINICAL TRIAL: NCT03938298
Title: Substudy of Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (ESTxENDS): Pulmonary Function Substudy (PulmENDS)
Brief Title: The ESTxENDS Trial: Pulmonary Function Substudy
Acronym: PulmENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss National Science Foundation (Other); Bernese Lung League (Unknown); Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332h
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Pulmonary Disease
MeSH Terms: conditions — Smoking Cessation; Lung Diseases

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ENDS (vaporizer/e-cig) and smoking cessation counseling
- Control group (Active Comparator)
  Interventions: Other: Smoking cessation counseling

INTERVENTIONS:
Other: ENDS (vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive standards of care, i.e. smoking cessation counseling and encouragement to use NRT. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date and again at week 1, 2, 4 and 8 after the target quit date. All participants will be followed over a 6-month period. After 6 months, participants will be asked to come to a final clinical visit.
  PFT and MBW will be performed at baseline and after the 6 months follow-up period in all participants of the substudy.
  Arms: Intervention group
Other: Smoking cessation counseling — Participants in the control group will receive standard of care only, i.e. i.e. smoking cessation counseling and encouragement to use NRT. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date and again at week 1, 2, 4 and 8 after the target quit date. All participants will be followed over a 6-month period. After 6 months, participants will be asked to come to a final clinical visit.
  PFT and MBW will be performed at baseline and after the 6 months follow-up period in all participants of the substudy.
  Arms: Control group

SUMMARY:
--> This is a substudy of the main ESTxENDS trial (NCT03589989). Pulmonary function outcomes should be considered secondary outcomes of the main smoking cessation outcome formulated in NCT03589989.

Cigarette smoking is the leading cause of preventable death in Switzerland and still more than a quarter of the Swiss population smokes cigarettes. Recently, electronic nicotine delivery systems (ENDS; also called vaporizer, e-cigarette or electronic cigarette) have become popular with smokers who want to stop smoking or reduce their exposure to inhaled chemicals since ENDS use appears to be safer than tobacco smoking. The inhaled ENDS aerosol appears safe in laboratory conditions, its long-term effects on pulmonary function remains unknown. This study will therefore investigate the impact of ENDS on lung function in smokers, who attempt to quit using ENDS compared with smokers, receiving only smoking cessation counseling with nicotine replacement therapy (NRT).

Multiple breath washout (MBW) is an established technique for assessment of peripheral airway function in pediatrics and its use is emerging in adult medicine, as it offers a better sensitivity to assess small airway disease before large airway involvement can be detected using conventional pulmonary function tests (PFT - spirometry, body plethysmography and diffusing capacity test). Preliminary evidence from limited studies suggest MBW parameters (LCI, Scond, Sacin) can be impaired in smokers with normal lung function and improve after smoking abstinence.

Primary objective of this substudy is to assess changes in LCI from baseline to 6 months post target quit date (TQD) in cigarette smokers randomized to the intervention group compared to the control group.

For the main ESTxENDS trial (NCT03589989), cigarette smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive standard of care, i.e. smoking cessation counseling and encouragement to use NRT. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date and again at week 1, 2, 4 and 8 after the target quit date. Participants in the control group will receive only standard of care. All participants will be followed over a 6-month period. After 6 months, participants will be asked to come to a final clinical visit.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion Criteria:

* Known hypersensitivity or allergy to contents of the e-liquid
* Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the scheduled study intervention, i.e. within the first 6-months of the study
* Persons having used ENDS or tobacco heating systems regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other medications with demonstrated efficacy as an aid for smoking cessation such as varenicline or bupropion within the 3 months preceding the baseline visit
* Persons who cannot attend the 6-month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in Lung Clearance Index (LCI) | Change from baseline to 6 months post quit date
  Measured by multiple breath washout (MBW) of a tracer gas (N2). LCI is defined as the cumulative expired volume/functional residual capacity (CEV/FRC) at 5% and 2.5% tracer gas concentration in the exhaled breath. An LCI with a z-score < + 1.645 (upper limit of normal according to Singer F et al, PLoS One. 2012;7(4):e36083) is considered normal.

SECONDARY OUTCOMES:
Lung Clearance Index (LCI) | 6 months post quit date
  Measured by multiple breath washout (MBW) of a tracer gas (N2). LCI is defined as the cumulative expired volume/functional residual capacity (CEV/FRC) at 5% and 2.5% tracer gas concentration in the exhaled breath. An LCI with a z-score < + 1.645 (upper limit of normal according to Singer F et al, PLoS One. 2012;7(4):e36083) is considered normal.
Changes in Scond and Sacin | Change from baseline to 6 months post quit date
  Measured by multiple breath washout (MBW). MBW assesses ventilation of the peripheral airways.
Scond and Sacin | 6 months post quit date
  Measured by multiple breath washout (MBW). MBW assesses ventilation of the peripheral airways.
Forced Expiratory Volume in 1 Second (FEV1) | 6 months post quit date
  Measured by spirometry. Spirometry is a conventional pulmonary function test measuring airflow.
Changes in Forced Expiratory Volume in 1 Second (FEV1) | Change from baseline to 6 months post quit date
  Measured by spirometry. Spirometry is a conventional pulmonary function test measuring airflow.
Forced Expiratory Volume in 1 Second/Functional Vital Capacity Ratio (FEV1/FVC) | 6 months post quit date
  Measured by spirometry. Spirometry is a conventional pulmonary function test measuring airflow.
Changes in Forced Expiratory Volume in 1 Second/Functional Vital Capacity Ratio (FEV1/FVC) | Change from baseline to 6 months post quit date
  Measured by spirometry. Spirometry is a conventional pulmonary function test measuring airflow.
Total Lung Capacity (TLC) | 6 months post quit date
  Measured by body plethysmography. Body plethysmography is a conventional pulmonary function test measuring lung volumes.
Changes in Total Lung Capacity (TLC) | Change from baseline to 6 months post quit date
  Measured by body plethysmography. Body plethysmography is a conventional pulmonary function test measuring lung volumes.
Residual Volume (RV) | 6 months post quit date
  Measured by body plethysmography. Body plethysmography is a conventional pulmonary function test measuring lung volumes.
Changes in Residual Volume (RV) | Change from baseline to 6 months post quit date
  Measured by body plethysmography. Body plethysmography is a conventional pulmonary function test measuring lung volumes.
Residual Volume to Total Lung Capacity (RV/TLC) | 6 months post quit date
  Measured by body plethysmography. Body plethysmography is a conventional pulmonary function test measuring lung volumes.
Changes in Residual Volume to Total Lung Capacity (RV/TLC) | Change from baseline to 6 months post quit date
  Measured by body plethysmography. Body plethysmography is a conventional pulmonary function test measuring lung volumes.
Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) | 6 months post quit date
  Measured by diffusing capacity test.
Changes in Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) | Change from baseline to 6 months post quit date
  Measured by diffusing capacity test.
Fraction of exhaled nitric oxide (FeNO) | 6 months post quit date
  Measured by the levels of nitric oxide in the exhaled breath.
Changes in Fraction of exhaled nitric oxide (FeNO) | Change from baseline to 6 months post quit date
  Measured by the levels of nitric oxide in the exhaled breath.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med, Study Director — Berner Institut für Hausarztmedizin; Universität Bern; Manuela Funke-Chambour, PD Dr. med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Switzerland (2):
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Department of Pneumology, Bern

REFERENCES:
- [Background] Farsalinos KE, Polosa R. Safety evaluation and risk assessment of electronic cigarettes as tobacco cigarette substitutes: a systematic review. Ther Adv Drug Saf. 2014 Apr;5(2):67-86. doi: 10.1177/2042098614524430. PMID 25083263
- [Background] Subbarao P, Milla C, Aurora P, Davies JC, Davis SD, Hall GL, Heltshe S, Latzin P, Lindblad A, Pittman JE, Robinson PD, Rosenfeld M, Singer F, Starner TD, Ratjen F, Morgan W. Multiple-Breath Washout as a Lung Function Test in Cystic Fibrosis. A Cystic Fibrosis Foundation Workshop Report. Ann Am Thorac Soc. 2015 Jun;12(6):932-9. doi: 10.1513/AnnalsATS.201501-021FR. PMID 26075554
- [Background] Robinson PD, Latzin P, Verbanck S, Hall GL, Horsley A, Gappa M, Thamrin C, Arets HG, Aurora P, Fuchs SI, King GG, Lum S, Macleod K, Paiva M, Pillow JJ, Ranganathan S, Ratjen F, Singer F, Sonnappa S, Stocks J, Subbarao P, Thompson BR, Gustafsson PM. Consensus statement for inert gas washout measurement using multiple- and single- breath tests. Eur Respir J. 2013 Mar;41(3):507-22. doi: 10.1183/09031936.00069712. Epub 2013 Feb 8. PMID 23397305
- [Background] Jetmalani K, Thamrin C, Farah CS, Bertolin A, Chapman DG, Berend N, Salome CM, King GG. Peripheral airway dysfunction and relationship with symptoms in smokers with preserved spirometry. Respirology. 2018 May;23(5):512-518. doi: 10.1111/resp.13215. Epub 2017 Nov 15. PMID 29141272
- [Background] Verbanck S, Schuermans D, Meysman M, Paiva M, Vincken W. Noninvasive assessment of airway alterations in smokers: the small airways revisited. Am J Respir Crit Care Med. 2004 Aug 15;170(4):414-9. doi: 10.1164/rccm.200401-037OC. Epub 2004 May 6. PMID 15130906
- [Background] Verbanck S, Schuermans D, Paiva M, Meysman M, Vincken W. Small airway function improvement after smoking cessation in smokers without airway obstruction. Am J Respir Crit Care Med. 2006 Oct 15;174(8):853-7. doi: 10.1164/rccm.200603-422OC. Epub 2006 Jun 23. PMID 16799076
- [Background] Singer F, Houltz B, Latzin P, Robinson P, Gustafsson P. A realistic validation study of a new nitrogen multiple-breath washout system. PLoS One. 2012;7(4):e36083. doi: 10.1371/journal.pone.0036083. Epub 2012 Apr 27. PMID 22558338